CLINICAL TRIAL: NCT00659360
Title: A Phase 2 Study of AZD0530 in Recurrent or Metastatic Soft Tissue Sarcoma
Brief Title: AZD0530 in Treating Patients With Recurrent Locally Advanced or Metastatic Soft Tissue Sarcoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-01054; PHL-054 (Other Grant/Funding Number: N01CM62203); CDR0000588034 (Other Grant/Funding Number: N01CM62203); PMH-PHL-054 (Other Grant/Funding Number: N01CM62203); N01CM62203 (NIH)
Record Dates: First submitted 2008-04-15; First posted 2008-04-16 (Estimated); Results first posted 2015-07-30 (Estimated); Last update posted 2018-06-29 (Actual); Status verified 2018-05

CONDITIONS: Adult Fibrosarcoma; Adult Leiomyosarcoma; Adult Liposarcoma; Adult Malignant Fibrous Histiocytoma; Adult Rhabdomyosarcoma; Dermatofibrosarcoma Protuberans; Endometrial Stromal Sarcoma; Recurrent Adult Soft Tissue Sarcoma; Recurrent Uterine Sarcoma; Stage III Adult Soft Tissue Sarcoma; Stage III Uterine Sarcoma; Stage IV Adult Soft Tissue Sarcoma; Stage IV Uterine Sarcoma; Uterine Carcinosarcoma; Uterine Leiomyosarcoma
MeSH Terms: conditions — Fibrosarcoma; Leiomyosarcoma; Liposarcoma; Histiocytoma, Malignant Fibrous; Rhabdomyosarcoma; Dermatofibrosarcoma; Sarcoma, Endometrial Stromal; Sarcoma | interventions — saracatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Arm I (Experimental): Patients receive oral AZD0530 (saracatinib ) at a dose of 175 mg, once daily, in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: saracatinib

INTERVENTIONS:
Drug: saracatinib — Given orally
  Other Names: AZD0530

SUMMARY:
This phase II trial is studying how well AZD0530 works in treating patients with recurrent locally advanced, or metastatic soft tissue sarcoma. AZD0530 may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
OBJECTIVES:

I. To assess the efficacy of AZD0530, in terms of disease control rate (i.e., response rate and stable disease rate), in patients with recurrent locally advanced or metastatic soft tissue sarcoma.

II. To assess the toxicity, time to progression, and response duration of AZD0530 in these patients.

OUTLINE: This is a multicenter study.

Patients receive oral AZD0530 once daily in the absence of disease progression or unacceptable toxicity.

After completion of study therapy, patients are followed every 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Leukocytes >= 3,000/mcL
* Histologically or cytologically confirmed soft tissue sarcoma including, but not limited to any of:

  * Malignant fibrous histiocytoma
  * Fibrosarcoma - non infantile
  * Leiomyosarcoma - not uterine
  * Liposarcoma
  * Non-rhabdomyosarcoma soft tissue sarcoma
  * Rhabdomyosarcoma, not otherwise specified
  * Carcinosarcoma of the uterus
  * Dermatofibrosarcoma
  * Endometrial stromal sarcoma
  * Leiomyosarcoma - uterus
* Recurrent or locally advanced or metastatic disease

  * No more than two prior lines of chemotherapy for metastatic disease (not including adjuvant chemotherapy)
* Measurable disease, defined as >= 1 unidimensionally measurable lesion >= 20 mm by conventional techniques or >= 10 mm by spiral CT scan

  * Target measurable lesion must not have been in previous radiation portal, unless progression of this lesion after radiotherapy has been documented
* ECOG performance status (PS) 0-2 or Karnofsky PS 60-100%
* Life expectancy > 12 weeks
* Recovered from all prior therapy
* Platelet count >= 100,000/mcL
* Hemoglobin > 9 g/dL
* Total bilirubin =< 1.25 times upper limit of normal (ULN)
* AST and ALT =< 3 times ULN
* Creatinine =< 1.5 times ULN OR creatinine clearance >= 50 mL/min
* Urine protein:creatinine ratio =< 1.0 OR 24-hour urine protein < 1,000 mg
* ANC >1,500/mcL
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 8 weeks after completion of study therapy
* No history of allergic reactions attributed to compounds of similar chemical or biological composition to AZD0530
* No QTc prolongation (defined as a QTc interval >= to 460 msecs) or other significant ECG abnormalities
* No poorly controlled hypertension (i.e., systolic blood pressure (BP) >= 140 mm Hg, or diastolic BP >= 90 mm Hg)
* No condition that impairs a patient's ability to swallow AZD0530 tablets, including any of the following:

  * Gastrointestinal tract disease resulting in an inability to take oral medication or a requirement for IV alimentation
  * Prior surgical procedures affecting absorption
  * Active peptic ulcer disease

Exclusion Criteria:

* At least 4 weeks since prior chemotherapy (6 weeks for nitrosoureas or mitomycin C)
* No intercurrent cardiac dysfunction including, but not limited to, any of the following:

  * Symptomatic congestive heart failure
  * Unstable angina pectoris
  * Cardiac arrhythmia
* No history of ischemic heart disease, including myocardial infarction
* No uncontrolled intercurrent illness including, but not limited to ongoing or active infection or psychiatric illness/social situations that would limit compliance with study requirements
* More than 4 weeks since prior radiotherapy
* More than 7 days since prior and no concurrent prohibited CYP3A4-active agents or substances
* No other concurrent investigational agents or commercial agents or therapies
* No concurrent combination antiretroviral therapy for HIV-positive patients
* No known brain metastases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2008-02; Primary Completion 2009-01 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Margaret von Mehren, Principal Investigator — University Health Network-Princess Margaret Hospital
Locations (4):
- Fox Chase Cancer Center, Rockledge, Pennsylvania, United States
- Canada (3):
  - Cross Cancer Institute, Edmonton, Alberta
  - University Health Network-Princess Margaret Hospital, Toronto, Ontario
  - Montreal General Hospital, Montreal, Quebec

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm I AZD0530: Patients receive oral AZD0530 once daily in the absence of disease progression or unacceptable toxicity.
  saracatinib: Given orally
Period: Overall Study
Arm/Group | Arm I AZD0530
Started | 17
Completed | 17
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Arm I: Patients receive oral AZD0530 once daily in the absence of disease progression or unacceptable toxicity.
  saracatinib: Given orally
Arm/Group | Arm I
Number analyzed (Participants) | 17
Age, Continuous [Median (Full Range); unit: years] | 65 [22 to 79]
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 8
  >=65 years | 9
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 6
Region of Enrollment [Number; unit: participants]
  United States | 8
  Canada | 9

OUTCOME MEASURES:

1. Primary Outcome: Disease Control Rate, Defined as the Number of Patients Who Achieved Complete Response, Partial Response or Stable Disease For a Period of More Than 4 Months.
Description: Response and progression will be evaluated using the new international criteria proposed by the Response Evaluation Criteria in Solid Tumors (RECIST) Changes in only the largest diameter (unidimensional measurement) of the tumor lesions; where CR is disappearance of all target lesions, PR is at least 30% decrease in the sum of longest diameter, PD is at least 20% increase in the sum of longest diameter recorded since the treatment started and SD is neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD
Time Frame: Up to 5 years
Measure: Number; unit: participants
Arm/Group | Arm I
Number analyzed (Participants) | 17
participants | 0

2. Secondary Outcome: Objective Response Rate
Description: Complete Response (CR) - Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions
Time Frame: Up to 5 years
Measure: Number; unit: participants
Arm/Group | Arm I
Number analyzed (Participants) | 17
participants | 0

3. Secondary Outcome: Overall Survival
Description: Median was estimated. The Kaplan-Meier method will be used to estimate overall survival estimates.
Time Frame: Up to 5 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm I
Number analyzed (Participants) | 17
months | 16.1 [3.8 to 17.9]

4. Secondary Outcome: Stable Disease Rate
Description: Achieved stable disease as their best response
Time Frame: Up to 5 years
Measure: Number; unit: participants
Arm/Group | Arm I
Number analyzed (Participants) | 17
participants | 2

5. Secondary Outcome: Duration of Response
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions;
  Objective Tumor Response "of more than 4 months" was counted toward the Disease Control Rate.
Time Frame: Up to 5 years
Population: Patients who had partial response, complete response or stable disease
Measure: Number; unit: participants
Arm/Group | Arm I AZD0530
Number analyzed (Participants) | 17
participants | 0

6. Secondary Outcome: Time to Disease Progression
Description: The Kaplan-Meier method will be used to estimate time to progression estimates.
  Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: Up to 5 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm I
Number analyzed (Participants) | 17
months | 1.7 [1.6 to 3.5]

ADVERSE EVENTS:
Arm/Group | Arm I
Serious Adverse Events (participants affected / at risk) | 5/17
Other Adverse Events (participants affected / at risk) | 17/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (N=17)
Hypokalemia (Metabolism and nutrition disorders) | 1
Proteinuria (Renal and urinary disorders) | 1
Lymphocyte count decreased (Investigations) | 2
Aspartate aminotransferase increased (Investigations) | 1
Fever (General disorders) | 2
Blood bilirubin increased (Investigations) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory, thoracic and mediastinal disorders - Other, specify - unspecified (Respiratory, thoracic and mediastinal disorders) | 2
Anemia (Blood and lymphatic system disorders) | 2
Fatigue (General disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (N=17)
Fatigue (General disorders) | 13
Anemia (Blood and lymphatic system disorders) | 12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less